CLINICAL TRIAL: NCT06647355
Title: Predicting Body Pain by Postural Related Problems in Middle-age and Older Adults Using Machine Learning
Brief Title: Evaluation of the Effect of a Clinical Exercise Programme on Plantar Distribution and Correction of Postural Asymmetries
Status: Completed | Type: Observational
Sponsor: University of Beira Interior (Other)
Responsible Party: Principal Investigator, Svitlana Dikhtyarenko, PhD Student, Principal Investigador, University of Beira Interior
Other Study IDs: CE-UBI-Pj-2023-030
Record Dates: First submitted 2024-10-06; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: This Study Highlights Differences in Baropodometry Between Genders
Keywords: Baropodometry, Bioimpedance, Artificial Intelligence

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- I: The 'M' point is on the heels of both feet.
  Interventions: Other: Effectiveness of physical exercise in preventing pain and improving plantar pressure distribution
- II: The 'M' point is located on the heel of the left foot and the forefoot of the right foot.
  Interventions: Other: Effectiveness of physical exercise in preventing pain and improving plantar pressure distribution
- III: Point 'M' is located on the heel of the right foot and the forefoot of the left foot.
  Interventions: Other: Effectiveness of physical exercise in preventing pain and improving plantar pressure distribution
- IV: The point of maximum pressure is in the forefoot area of both feet.
  Interventions: Other: Effectiveness of physical exercise in preventing pain and improving plantar pressure distribution
- V: The 'M' point is in the medial zone on both feet.
  Interventions: Other: Effectiveness of physical exercise in preventing pain and improving plantar pressure distribution
- VI: The 'M' point is located on the left midfoot and right rearfoot.
  Interventions: Other: Effectiveness of physical exercise in preventing pain and improving plantar pressure distribution
- VII: The 'M' point is located on the right midfoot and left rearfoot.
  Interventions: Other: Effectiveness of physical exercise in preventing pain and improving plantar pressure distribution

INTERVENTIONS:
Other: Effectiveness of physical exercise in preventing pain and improving plantar pressure distribution — At the beginning of the study, the participants underwent a baropodometric and photometric analysis. At the same time, anthropometric data and self-assessed body pain data were collected. For 12 continuous weeks, the participants completed a training programme that included specific exercises designed for each group. At the end, the baropodometry images were analysed again, which led to the final conclusion of the study.

SUMMARY:
The aim of this study was to identify significant variables that contribute to the association between postural problems, plantar pressure distribution and levels of bodily pain in middle-aged and elderly adults. The researchers' hypothesis is that plantar pressure characteristics and postural asymmetries differ according to gender, are related to body composition and predict pain levels. The study described here is the only one to include variables that make it possible to identify body asymmetries in a postural analysis, based on the distribution of plantar pressure and body composition.

DETAILED DESCRIPTION:
The study employed an observational cross-sectional design. A convenience sample was recruited to analyse differences between men and women in anthropometrics, body composition, plantar pressure distribution, and pain levels. Without intervention, researchers observed and recorded data at a single time point, allowing comparisons between sexes and exploring correlations among the measured variables. This type of design allowed a snapshot view of the differences and associations present within the sample.

ELIGIBILITY:
Inclusion criteria:

* Participants had to be at least eighteen years old and physically fit. All participants had to complete the PAR-Q (health questionnaire), psychological well-being questionnaire (EBEP) and sign the free, informed and informed consent form (CLIE).

Exclusion criteria:

* In order to reduce the risk of injury or aggravation of known diseases, the researchers chose the following exclusion criteria: serious orthopaedic problems (prosthesis fitting, recent orthopaedic surgery), reported neurological problems (requiring daily medication), cardiopulmonary diseases (pacemaker, use of oxygen cylinders) and pregnant women.

Ages: 18 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of the present study consisted of 52 (n=52) participants of both sexes. The majority of study participants were female, comprising 67.3% (n=35), while 32.7 % of the sample were male (n=17). The mean age of participants was 57.35 years in males and 64.69 years in females.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Importance and benefits of physical exercise in preventing pain and improving quality of life | 12 weeks
  Sequencing of the training plan

SECONDARY OUTCOMES:
Bodily pain and discomfort | 12 weeks
  Relationship between posture and pain

OTHER OUTCOMES:
Significant changes in baropodometry images | 12 weeks
  Physical exercise and changes in footsteps

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Mr Forte, PhD, Study Director — University of Beira Interior; Dulce Ms Esteves, PhD, Study Director — University os Beira Interior
Locations (1):
- Svitlana Dikhtyarenko, Setúbal, Rua Das Areias, 11 - 2, Portugal

IPD SHARING:
Plan to Share IPD: No